CLINICAL TRIAL: NCT07254637
Title: Randomized, Double-blind, Multicentre Trial of Tocilizumab Versus Placebo in Chronic Polyarticular Inflammatory of Calcium Pyrophosphate Deposition Disease Refractory to Standard Treatments
Brief Title: Tocilizumab in Chronic Inflammatory CPPD Disease
Acronym: TociCCAre
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fresenius AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP220790
Record Dates: First submitted 2025-08-14; First posted 2025-11-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Calcium Pyrophosphate Deposition Disease
MeSH Terms: conditions — Chondrocalcinosis | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: TociCCAre is a phase II, randomised, double-blind, placebo-controlled comparative study. The study aims to demonstrate the efficacy of tocilizumab in treating chronic polyarticular inflammation associated with CPP crystals.
  It is a superiority study with 1:1 randomisation into two parallel groups.
  This multicentre study has 12 participating centres, including centres specialising in microcrystalline diseases and a reference centre for Gitelman syndrome (one of whose complications is extensive PPC crystal deposition), located at the HEGP hospital in Paris.
  Patients will be enrolled during consultations and hospitalisations by the principal investigator or their co-investigators.
Who Masked: Participant
Masking Description: Pharmacy Process: Upon email notification, the pharmacy prepares and dispenses the tocilizumab or placebo. If unable to reconstitute it, they provide a nominative patient kit for external reconstitution.
  Non-protocol Handlers: Specially trained nurses reconstitute treatment bags discreetly. Each center has a designated trainer to build a team of these off-protocol handlers.
  Pharmacy Oversight: The hospital pharmacist ensures proper management of investigational products. Compliance is checked by a CRA during monitoring.
  Blinding Strategy:
  A blind CRA monitors clinical activities. An open CRA manages pharmacy stock and is aware of treatment allocation. The trial is double-blind to prevent bias for both patients and investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab, 8 mg/kg/month, IV infusion for 3 months
  Tocilizumab, an anti-IL-6R monoclonal antibody, was approved in January 2009 for the treatment of rheumatoid arthritis. Its indications have since been extended, particularly for the treatment of giant cell arteritis, juvenile chronic arthritis, and severe cytokine release syndrome induced by chimeric antigen receptor T-cell (CAR-T) therapy.
  Arms: Tocilizumab
Other: Placebo — Saline placebo, IV infusion / month for 3 months
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to determine the efficacy of tocilizumab (an IL-6 inhibitor) in treatment-refractory chronic inflammatory forms of CPPD.

The main questions this trial aims to answer are:

* Can tocilizumab improve joint pain in patients with chronic inflammatory CPPD disease?
* Does tocilizumab improve quality of life in patients with chronic inflammatory CPPD disease?

Participants will receive a monthly infusion of tocilizumab or placebo for three months.

DETAILED DESCRIPTION:
Calcium pyrophosphate deposition (CPPD) disease affects 4 to 7% of the adult population. CPP crystals are responsible for inflammatory flares affecting one or more joints. The inflammation triggered by CPP crystals resembles that associated with sodium urate crystals in gout and depends on inflammatory cytokines such as interleukins (IL-) 1β and -6. The usual treatments are those used in gout flares (colchicine, NSAIDs, corticosteroids, IL-1β inhibitors), and most often control monoarticular involvement. The chronic inflammatory polyarticular form, on the other hand, is more difficult to treat, causing significant pain and disability, as well as joint destruction. In refractory forms, or in cases of intolerance to standard treatments, alternative therapies are required. In this context, the investigators treated 11 patients with refractory chronic inflammatory CPPD with tocilizumab (TCZ), an anti-IL-6 receptor (IL-6R) monoclonal antibody. After 3 monthly infusions, improvement was estimated at over 75% (PMID 2213498). Our hypothesis is that inhibiting IL-6 is an effective therapeutic option in chronic inflammatory CPPD refractory to conventional therapies.

Main objective and primary endpoint:

* To demonstrate the efficacy of IL-6 inhibition in treatment-refractory chronic inflammatory forms of CPPD disease.
* Our endpoint will be the change in global pain VAS between initiation and M4, i.e. one month after the 3rd infusion. VAS will be assessed after 24 hours off analgesics.

Secondary objectives and endpoints:

* Efficacy: DAS44, number of swollen, painful joints, overall disease activity VAS, fatigue VAS; overall effect on pain: area under the VAS curve (AUC); proportion of patients responding from M2 to M6 (improvement ≥ 50% of initial pain VAS) and complete response (improvement ≥ 80% of initial pain VAS); relapse rate; improvement in quality of life (SF-36, HAQ, EQ-5D-3L questionnaires)
* Tolerance: infusion reactions, infections, neutropenia, hepatic cytolysis, lipid profile

This is a phase III, multicentre, randomized, controlled, double-blind, superiority study, including 2 parallel groups with a 1:1 distribution. This trial will involve adults suffering from the chronic inflammatory polyarticular form of CPPD disease.

This study will involve 80 participants recruited in 12 centres in France.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Diagnosis of CPPD according to ACR/EULAR 2023 classification criteria
* Persistent inflammatory pain (> 3 months) or ≥ 2 arthritics/month
* Number of painful joints (NAD) > 3
* Overall pain VAS (0_100) > 40 mm
* Failure, intolerance or impossibility of repeated use of usual treatments: colchicine, NSAIDs, corticosteroids and anakinra
* Use of an effective method of contraception in women of childbearing age until 3 months after the end of the study.
* Informed consent

Exclusion Criteria:

* Presence of anti-CPP antibodies > 50 IU/ml
* Recurrent or chronic infections
* History of severe infection (= requiring hospitalization)
* Active infection
* Vaccination with live or attenuated vaccine within 4 weeks prior to inclusion
* History of intestinal ulceration or diverticulitis Untreated latent tuberculosis
* History of viral hepatitis B ou C
* Symptoms suggestive of demyelinating disease of the central nervous system
* History of cancer, active cancer, or suspected cancer
* Neutropenia < 2000 elements/mm3, thrombocytopenia < 100 000/mm3
* Elevated transaminases > 3 x ULN
* Known hypersensitivity to the active substance or one of the excipients;
* Known severe immune deficiency
* Patients not meeting classification criteria
* Concomitant treatment with biological or targeted therapies, or immunosuppressive therapy (including methotrexate, leflunomide, azathioprine), systemic corticosteroids, anakinra, IL-6 inhibitors in subcutaneous injection, anti-TNF agents, and JAK. If these treatments are used before inclusion, a washout period corresponding to at least five times their respective mean terminal half-life must be respected.
* inhibitors.
* Previous treatment with tocilizumab
* Concomitant treatment with methylprednisolone, dexamethasone, atorvastatin, calcium channel blockers, theophylline, warfarin, phenprocoumon, phenytoin, cyclosporine or benzodiazepines
* Dyslipidemia, hypertension or poorly controlled cardiovascular disease
* Scheduled surgery
* Difficulty to understand French, illiteracy
* Pregnant women, women in labor or nursing mothers
* Persons deprived of their liberty, adults under legal protection or unable to express their consent
* Persons not affiliated to a social security scheme or beneficiaries of such a scheme
* Participation in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Change in overall pain VAS | 6 months
  Overall pain will be assessed, after 24 hours of discontinuation of analgesics, using a visual analogue scale (VAS) ranging from 0 (no pain) to 100 mm (worst pain ever experienced), at inclusion, before each infusion at months M1, M2, M3, then at M4 (primary outcome) and M6.

SECONDARY OUTCOMES:
Change in the number of swollen and tender joints | 6 months
  Disease Activity Score (DAS44), number of swollen and painful joints, Patient assessment of overall disease activity by a visual analogue scale (VAS) ranging from 0 (no activity) to 100 mm (maximal activity). Those outcomes will be assessed at inclusion, before each infusion at months M1, M2, M3, then at M4 (primary outcome) and M6
Overall effect on pain | 6 months
  Area under the curve (AUC) of the overall pain visual analogue scale (VAS) ranging from 0 (no pain) to 100 mm (worst pain ever experienced) based on assessments at baseline, before each infusion at months M1, M2, M3 and at M4 and M6 (end of the study). Overall pain VAS will be collected after a 24-hour washout of analgesics.
Response to treatment / relapse | 6 months
  Response to treatment will be defined as an improvement ≥ 50% of initial pain visual analogue scale (VAS) ranging from 0 (no pain) to 100 mm (worst pain ever experienced) Complete response will be defined as an improvement ≥ 80% of initial pain VAS This outcome will be assessed from M2 to M6.
  Relapse will be assessed in responders at 6 months, and the time from response to relapse will be determined.
Flares (ESR) | 6 months
  Outcome Measures - Inflammatory Biomarkers
  Erythrocyte Sedimentation Rate (ESR) Unit: millimeters (mm) Frequency: measured at each visit
  No aggregation of this measure is planned to produce a composite value. If aggregation is considered (e.g., to generate an overall inflammation score), a validated statistical method will be specified.
Flares (CRP) | 6 months
  Outcome Measures - Inflammatory Biomarkers
  C-reactive Protein (CRP) Unit: milligrams per liter (mg/L) Frequency: measured at each visit
  No aggregation of this measure is planned to produce a composite value. If aggregation is considered (e.g., to generate an overall inflammation score), a validated statistical method will be specified.
Flares (IL-6) | 6 months
  Outcome Measures - Inflammatory Biomarkers
  Interleukin-6 (IL-6) Unit: picograms per milliliter (pg/mL) Frequency: measured at each visit
  No aggregation of this measure is planned to produce a composite value. If aggregation is considered (e.g., to generate an overall inflammation score), a validated statistical method will be specified.
Quality of life's Questionnaires (SF-36) | 6 months
  Full Title: Short Form 36 Health Survey (SF-36) Scale Range: 0 to 100 per subscale Interpretation: Higher scores indicate better health status or quality of life Time Points: Baseline, prior to each infusion, and at Months 4 and 6 (M4 and M6) Unit: Score
  This questionnaire will be analyzed and reported as a distinct outcome measure, in accordance with its specific scoring system.
Quality of life's Questionnaires (HAQ) | 6 months
  Full Title: Health Assessment Questionnaire (HAQ) Scale Range: 0 to 3 Interpretation: Higher scores indicate worse functional ability (i.e., more disability) Time Points: Baseline, prior to each infusion, and at Months 4 and 6 (M4 and M6) Unit: Score
  This questionnaire will be analyzed and reported as a distinct outcome measure, in accordance with its specific scoring system.
Quality of life's Questionnaires (EQ-5D-3L) | 6 months
  Full Title: EuroQol Five Dimensions Three Levels (EQ-5D-3L) Scale Range: 0 to 100 Interpretation: Higher scores indicate better health-related quality of life Time Points: Baseline, prior to each infusion, and at Months 4 and 6 (M4 and M6) Unit: Index value
  This questionnaire will be analyzed and reported as a distinct outcome measure, in accordance with its specific scoring system.
Patient Safety - Number of Participants with Adverse Events | 6 months
  Outcome Measure - Number of Participants with Adverse Events
  Description: Number of participants experiencing any of the following safety-related events at each visit:
  * Infusion reactions
  * Neutropenia
  * Thrombocytopenia
  * Hepatic cytolysis
  * Severe infections
  * Treatment-related adverse events
  * Abnormal changes in lipid profile
  Unit of Measure: Count (participants) Time Points: Each visit Note: Each event type will be recorded and analyzed separately but reported under a unified outcome measure to reflect overall safety.
Patient Safety - Number of patients with abnormal laboratory tests results - Mean Neutrophil Count | 6 months
  Description: Mean neutrophil count measured from blood samples collected at each visit.
  Unit of Measure: normal: 2500-8000/μL; AE: <1500/μL
Patient Safety - Number of patients with abnormal laboratory tests results - Mean Platelet Count | 6 months
  Description: Mean platelet count measured from blood samples collected at each visit.
  Unit of Measure: normal: 150,000-400,000/μL; AE: <75,000/μL
Patient Safety - Number of patients with abnormal laboratory tests results - Mean Transaminase Levels | 6 months
  Description: Mean levels of transaminases (e.g., ALT, AST) measured to assess hepatic cytolysis.
  Unit of Measure: ALT/AST normal: <40 U/L; AE: >3×ULN
Patient Safety - Number of patients with abnormal laboratory tests results - Mean Lipid Profile Values | 6 months
  Description: Mean values of lipid profile components (e.g., total cholesterol, LDL, HDL, triglycerides) measured at each visit.
  Unit of Measure: normal: TC <200, LDL <130, HDL >45/55, TG <150 mg/dL

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Groupe Hospitalier de l'Institut Catholique de Lille, Lomme, Lille
  - Lariboisière hospital, Paris, Paris Paris
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes, Paris
  - CHU de Dijon, Dijon
  - CHU de Nantes, Nantes
  - Hôpital Bichat Claude-Bernard, Paris
  - Hôpital de la Croix Saint-Simon, Paris
  - Hôpital Tenon, Paris
  - Groupe Hospitalier Intercommunal Le Raincy-Montfermeil, Paris
  - Hôpital Le Kremlin Bicêtre, Paris
  - CHU de Rennes, Rennes
  - CHU de Saint-Étienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No